CLINICAL TRIAL: NCT04842097
Title: Online Mindfulness-based Stress Reduction Intervention for Chronic Pain in Individuals Waiting for Health Care Services: a Study Protocol for a Pilot Randomized Controlled Trial (RCT)
Brief Title: Online Mindfulness-based Stress Reduction Intervention for People With Chronic Pain Waiting for Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Diana Zidarov, site researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRIR-1499-1120/multi
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pain
Keywords: mindfulness-based stress reduction intervention
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: A two group parallel single blind pilot RCT
Who Masked: Investigator, Outcomes Assessor
Masking Description: It is not possible to blind the participants to group allocation due to the nature of the mindfulness-based stress reduction intervention; however, the outcome assessor, who will administer the outcome questionnaires to the participants will be blinded to the participants' group allocation as well the investigator and the data analyst who will conduct the analysis ensuring neutrality of the outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction intervention (Experimental): Online 8-week group program, once per week
  Interventions: Behavioral: Mindfulness-based stress reduction
- Waiting list (No Intervention): Controls will not receive any intervention during this time. They are on chronic pain clinics waiting list

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — An online mindfulness-based stress reduction intervention will be administered in a group format of maximum 15 participants, once a week for 120 minutes for 8 weeks by an experienced therapist trained in MBSR. Sessions will include sitting and lying meditation, hatha yoga and a body scan where attention is sequentially focused on different parts of the body. Individual autonomous practice between 30-45 minutes, 6 times / week will also be recommended. To support individual autonomous practice, a daily diary and two guided videos (around 35 minutes/each) were created.
  Arms: Mindfulness-based stress reduction intervention

SUMMARY:
The goal of this project is to explore the feasibility and the efficacy of a online mindfulness-based stress reduction intervention for people with chronic pain waiting for secondary or tertiary health care services

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-85
* Self-reported diagnosis of chronic non-cancer pain
* Chronic non-cancer pain duration of 3 months or more
* Chronic non-cancer pain experienced during 4 days or more per week
* Average pain intensity of 4 or more out of 10 in the last seven days
* French or English fluency
* Access to Wi-Fi
* Be able to attend a weekly two-hour MBSR virtual session for eight consecutive weeks

Exclusion Criteria:

* Cancer-related chronic pain
* Currently receiving or have received in the last 24 months coordinated care in pain clinics, hospitals or rehabilitation centers.
* Current or recent participation (in the last 12 months and more than 12 sessions) of cognitive-behavioral therapy or MBSR program
* Having an unstable psychological conditions such as depression, bipolar disorder, post-traumatic stress disorder, psychotic disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Participants retention rate | 2 months
  The percentage of participants who have completed the 8 online MBSR sessions
Participants participation rate | 12 months
  The percentage of participants on waiting lists who agreed to participate in the intervention

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Global-10 | Change from week start of MBSR intervention (week 0) to end of intervention (week 8), 3-month follow-up (week 21)
  Change in domains of health and functioning as measured by the PROMIS Global-10, score range is 7-35 with increases in scores meaning better outcome
Patient-Reported Outcomes Measurement Information System 29 | Change from week start of MBSR intervention (week 0) to end of intervention (week 8), 3-month follow-up (week 21)
  Change in 8 health-related quality of life domains as measured by the PROMIS 29. PROMIS-29 is a generic patient reported outcome measure, which includes four items from each of the seven PROMIS domains (physical function, depression, anxiety, fatigue, sleep disturbance, and ability to participate in social roles and activities, pain interference) and a single item on pain intensity. Each item has five response options (values 1 to 5), except for the pain intensity item which has eleven response options (values 0 to 10). A total raw score is computed for each domain as the sum of the response to each question within the domain, leading to seven domain scores, each from 4 to 20.
French-Canadian Chronic Pain Self-Efficacy Scale | Change from week start of MBSR intervention (week 0) to end of intervention (week 8), 3-month follow-up (week 21)
  The French-Canadian Chronic Pain Self-Efficacy Scale (Lacasse et al., 2015) is a 6-item scale that measures an individual's confidence in his/her ability to manage chronic pain in general and pain-related symptoms. Items are rated on a 10-point Likert scale ranging from 1 = not at all confident to 10 = entirely confident. Score range is 6-60 with higher scores reflecting greater chronic pain self-efficacy.
Chronic Pain Acceptance Questionnaire | Change from week start of MBSR intervention (week 0) to end of intervention (week 8), 3-month follow-up (week 21)
  The Chronic Pain Acceptance Questionnaire (CPAQ-8; Fish et al., 2010 ) is an 8-item scale comprised of two subscales: activity engagement and pain willingness. Items are scored on a 7-point Likert scale ranging from 0 = never true to 6 = always true. Score range is 0-48 with increases in scores meaning better outcome.
Global Rating of Change Scale | 3-month follow-up (week 21)
  The Global Change Rating Scale (11-point visual analogue scale raging from minus 5 to plus 5) will be used to assess the participants' perception of improvement (or decline) in relation to their self-efficacy in manging pain at the end of the MBSR intervention.
Pain Catastrophizing Scale | Change from week start of MBSR intervention (week 0) to end of intervention (week 8), 3-month follow-up (week 21)
  Change in pain catastrophizing as measured by the Pain Catastrophizing Scale (French Canadian version). PCS is a 13-item measure using a 5-point Likert scale (0=not at all, 4=all the time) with score range between 0-52 with decreases in scores meaning better outcome.
Pain Disability Index | Change from week start of MBSR intervention (week 0) to end of intervention (week 8), 3-month follow-up (week 21)
  Change in pain disability as measured by the The French-Canadian Pain Disability Index (score range is 0-70 with decreases in scores meaning better outcome)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Association québécoise de la douleur chronique, Montreal, Quebec
  - Centre de réadaptation Layton-Lethbridge-Mackay, Montreal, Quebec
  - Hôpital de Verdun, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No